CLINICAL TRIAL: NCT05724303
Title: The Effects of Integrative Neuromuscular Training on Physical Activity, Gait, Strength, and Body Composition in Overweight and Obese Children
Brief Title: The Effects of Integrative Neuromuscular Training on Physical Function in Overweight Children
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: St. Mary's University, Twickenham (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: StMarysUC8
Record Dates: First submitted 2022-12-15; First posted 2023-02-13 (Actual); Last update posted 2023-02-13 (Actual); Status verified 2023-02

CONDITIONS: Obesity; Childhood Obesity
MeSH Terms: conditions — Obesity; Pediatric Obesity

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Training group (Experimental): 8-week neuromuscular training program
  Interventions: Other: 8-week neuromuscular training program
- Control group (No Intervention)

INTERVENTIONS:
Other: 8-week neuromuscular training program — Training program consisting of two neuromuscular training sessions per week
  Arms: Training group

SUMMARY:
Childhood obesity is an ongoing and increasing issue, resulting in changes in body mass which cause biomechanical alterations in the lower limbs. Exercise interventions have been effectiveness at causing positive changes to the lower limbs gait, strength and functioning but children often report lack of enjoyment from the sessions which inhibits long term changes. This intervention takes a neuromuscular exercise approach whilst considering the psychological needs of children to motivate them to participate in the intervention and physical activity.

ELIGIBILITY:
Inclusion Criteria:

* children aged 8-11 years old
* overweight/obese children

Exclusion Criteria:

* children who have not given consent or had parental consent to participate
* children who fall outside of the selected age range
* children who have a physical or mental impairment that will affect their ability to participate in the procedures in the laboratory and intervention settings

Ages: 8 Years to 11 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 24 (Estimated)
Dates: Start 2023-02-24 (Estimated); Primary Completion 2024-06-28 (Estimated); Study Completion 2024-06-28 (Estimated)

PRIMARY OUTCOMES:
Change in body fat percentage | From baseline to end of 8-week training program and to end of 8-week follow-up
  Bioelectrical impedance analysis of fat mass relative to body mass
Change in fat free mass | From baseline to end of 8-week training program and to end of 8-week follow-up
  Bioelectrical impedance analysis of fat free mass relative to body mass
Change in body mass index (BMI) | From baseline to end of 8-week training program and to end of 8-week follow-up
  BMI calculated with height measured barefoot on weight scales and height measured barefoot on Stadiometer and Z-score based on standard measures for age and gender. A reduction in BMI is a positive change.
Change in Hip 3d gait analysis | From baseline to end of 8-week training program and to end of 8-week follow-up
  3D joint angle, moment and power waveforms during stance phase. Moment and power dimensionless and normalised to body mass and leg length. Time normalised to 100% of stance and walking at a self-selected pace.
Change in Knee 3d gait analysis | From baseline to end of 8-week training program and to end of 8-week follow-up
  3D joint angle, moment and power waveforms during stance phase. Moment and power dimensionless and normalised to body mass and leg length. Time normalised to 100% of stance and walking at a self-selected pace.
Change in Ankle 3d gait analysis | From baseline to end of 8-week training program and to end of 8-week follow-up
  3D joint angle, moment and power waveforms during stance phase. Moment and power dimensionless and normalised to body mass and leg length. Time normalised to 100% of stance and walking at a self-selected pace.
Change in Foot 3d gait analysis | From baseline to end of 8-week training program and to end of 8-week follow-up
  Angle of the forefoot, midfoot, rearfoot and shank during the stance phase when walking at a self-selected pace.
Change in lower limb strength relative to body mass | From baseline to end of 8-week training program and to end of 8-week follow-up
  Lower limb strength measured on Isokinetic Dynamometer in hip flexion/extension, hip abduction/adduction, knee flexion/extension, ankle plantarflexion/dorsiflexion. Maximal moments allometrically scaled to body mass
Change in lower limb strength relative to fat free mass | From baseline to end of 8-week training program and to end of 8-week follow-up
  Lower limb strength measured on Isokinetic Dynamometer in hip flexion/extension, hip abduction/adduction, knee flexion/extension, ankle plantarflexion/dorsiflexion. Maximal moments allometrically scaled to fat free mass
Change in physical functioning: six-minute timed walk | From baseline to end of 8-week training program and to end of 8-week follow-up
  Distance walked at a self-selected speed for six minutes
Change in physical functioning: sit-to-stand test | From baseline to end of 8-week training program and to end of 8-week follow-up
  The amount of repetitions of moving from a sitting position with knees at 90 degrees flexion to an upright standing position and return in one minute. Arms fixed across chest.
Change in physical functioning: timed up and go test | From baseline to end of 8-week training program and to end of 8-week follow-up
  Time taken to rise from a seated position with knees at 90 degrees flexion and arms across chest, walk 3m and return back to seated position
Change in physical functioning: single leg stand eyes open | From baseline to end of 8-week training program and to end of 8-week follow-up
  Maximal time to maintain balance on one leg with hands on hip and free leg bent to 90degrees flexion
Change in physical functioning: single leg stand eyed closed | From baseline to end of 8-week training program and to end of 8-week follow-up
  Maximal time to maintain balance on one leg with eyes closed, hands on hip and free leg bent to 90degrees flexion
Change in physical activity: percentage of time spent in sedentary activity levels | From baseline to end of 8-week training program and to end of 8-week follow-up
  Accelerometer data captured and time spent in sedentary level expressed as a percentage of time worn. Accelerometers worn on right side waist for one week.
Change in physical activity: percentage of time spent in moderate to vigorous activity levels | From baseline to end of 8-week training program and to end of 8-week follow-up
  Accelerometer data captured and time spent in moderate to vigorous level expressed as a percentage of time worn. Accelerometers worn on right side waist for one week.
Change in motivation towards physical activity | From baseline to end of 8-week training program and to end of 8-week follow-up
  Behavioural Regulation in Exercise Questionnaire to measure motivation towards physical activity

CONTACTS AND LOCATIONS:
Overall Officials: Ryan Mahaffey, PhD, Principal Investigator — St. Mary's University, Twickenham
Locations (1):
- Three Bridges, Ealing, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No